CLINICAL TRIAL: NCT00577785
Title: A Multi-Center Study to Obtain Full Thickness Bladder Tissue Specimen From Subjects Undergoing Cystectomy Surgery
Brief Title: Study to Obtain Full Thickness Bladder Tissue From Subjects Undergoing Cystectomy Surgery
Status: Completed | Type: Observational
Sponsor: Tengion (Industry)
Responsible Party: Sunita Sheth, MD Chief Medical Officer, Tengion, Inc
Other Study IDs: TNG-CL005
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-12

CONDITIONS: Cystectomy
Keywords: cystectomy
MeSH Terms: interventions — Tissue and Organ Procurement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cystectomy group: Subjects undergoing planned cystectomy who agree to provide bladder tissue from removed bladder post cystectomy and/or cystoscopic biopsy tissue prior to cystectomy
  Interventions: Other: tissue procurement

INTERVENTIONS:
Other: tissue procurement — No intervention. Tissue procurement study.

SUMMARY:
The objective of this study is to obtain bladder tissue specimens from patients otherwise undergoing cystectomy for use in research and training of personnel at Tengion, Inc.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 to 90 years and undergoing a cystectomy surgery
* Willing and able to give signed informed consent

Exclusion Criteria:

* Known active infection
* Known colonization with MRSA or VRE
* Receipt of blood or blood products for transfusion during the previous 3 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients otherwise undergoing cystectomy
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2007-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of bladder tissue from patients underogoing radical cystectomy | ongoing throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Sunita Sheth, MD, Study Director — Tengion, Inc
Locations (1):
- University of Southern California, Los Angeles, California, United States